CLINICAL TRIAL: NCT02504255
Title: Evaluation of Immunological Markers, Inflammatory and Clinical Relapse Psychological Predictive During Crohn's Disease : A Multicenter Cohort
Brief Title: Evaluation of Immunological Markers, Inflammatory and Clinical Relapse Psychological Predictive During Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2010.630
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Crohn Disease
Keywords: Crohn disease; inflammatory biomarkers; immunologic markers; calprotectin
MeSH Terms: conditions — Crohn Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Crohn's Disease: patients will have biological samplings (blood, urine and faecal sampling) and will fill questionnaires to assess their stress and adaptation
  Interventions: Biological: Biological samplings; Other: Questionnaires

INTERVENTIONS:
Biological: Biological samplings — Blood, urine and faecal sampling every 3 months
Other: Questionnaires — patients fill several questionnaires every month to assess stress and adaptation parameters

SUMMARY:
Crohn disease (CD) usually evolves by surges interspersed by periods of unpredictable remission. the probability of recurrence of CD in a patient in remission is even stronger if it pre-exists endoscopic lesions of the intestinal mucosa.

The mucosal healing exploration needs the realization of an ileo-colonoscopy under general anesthesia which is an invasive procedure, restrictive and expensive, thus prohibiting its too frequent repetition. we do not currently have noninvasive and reliable markers able to predict the occurrence of thrust of CD and allow the introduction of a more suitable treatment.

Indeed, relapse prevention is the best way to avoid complications and formation of lesions that lead to the irreversible medical treatment failure and surgery.

Since during the CD, it is the immunological changes that lead to inflammation and lesions, we make the assumption that the ability of certain markers immunological to predict a relapse of CD is higher than that of other in particular inflammatory markers.

This work should help to identify the profile of patients with CD in remission but at high risk of recurrence. It will specify i) the potential new markers immunological, from the pre-clinical research, predict the onset of a recurrence of CD ; ii) the predictive interest of different inflammatory markers used in routine or during the CD evaluation ; iii) Finally, the stress and the management of stressful events in the occurrence of a relapse.

This work also will specify the evolution of different markers at the moment of thrust

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years.
* Patient with CD previously diagnosed according to standard criteria.
* Patient remission (HBS≤4) for at least 3 months and has not received corticosteroids (including budesonide) in the 3 months before.
* Patient without concomitant treatment of Crohn's disease or as stable dose (5-ASA, corticosteroids, immunosuppressants, anti-TNF) immunosuppressants (azathioprine, Purinethol, methotrexate) and / or anti-TNF and / or 5- amino salicylates (5-ASA) for at least 6 months.
* Patient who signed a consent.
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* A patient with an active CD (HB score≥5).
* Patient who relapsed in the previous three months before inclusion.
* Patient who received corticosteroids (including budesonide) in the 6 months prior to inclusion.
* Patients on stable dose of non-anti-TNF in the 6 months prior to inclusion.
* Patient taking nonsteroidal anti-inflammatory drugs or antibiotics.
* Patient with complications of intestinal sub-occlusion type fistulas or abdominal abscesses.
* Patient with exclusive perianal disease or a predominate perianal manifestation.
* Pregnant women (examination).
* Patient who is the subject of extensive intestinal resection (> 1 m).
* Patient with ileostomy or colostomy.
* Patient on legal protection measure or who does not have the legal capacity to consent
* Lack of signed written consent of the patient.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn Disease
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Correlation between new immunological markers rate and Crohn's Disease relapse | within 15 months
  This outcome will help us to show that regular monitoring of new immunological markers (serum markers of cytotoxicity of lymphocytes, pro- and anti-inflammatory cytokines and urinary and fecal neopterin) let us predict relapse of the disease

SECONDARY OUTCOMES:
Correlation between usual immunological markers rate and Crohn's Disease relapse | within 15 months
  This outcome will help us to test the ability of inflammatory markers which are already routinely used for diagnostic purposes to predict relapse of CD. These "usual" markers are : fecal calprotectin and lactoferrin, serum ultrasensitive C-Reactive Protein (CRP) and erythrocyte sedimentation rate (ESR)) is being evaluated (serum S100A12 protein, fecal, alpha-1-glycoprotein (orosomucoid) alpha-2 globulin)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Hôpital Hôtel Dieu - Service d'Hépato-Gastroentérologie, Clermont-Ferrand
  - Hospices Civils de Lyon - Groupement Hospitalier Sud - Service d'Hépato-Gastroentérologie, Pierre-Bénite
  - CHU Hôpital Nord - Service d'Hépato-Gastroentérologie, Saint-Etienne